CLINICAL TRIAL: NCT01703182
Title: Transcutaneous Oximetry, Transcutaneous Carbon Dioxide and Supplemental Oxygen Therapy in Lower Limb Amputations - An Observational Study
Brief Title: Transcutaneous Oximetry, Transcutaneous Carbon Dioxide and Supplemental Oxygen Therapy in Lower Limb Amputations
Acronym: TCOM
Status: Terminated | Type: Observational
Why Stopped: Stopped due to feasibility
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Richard Whitlock, Assistant Professor, McMaster University
Organization: McMaster University (Other)
Other Study IDs: TCOM-2012
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Amputation Wound
Keywords: transcutaneous oximetry; transcutaneous carbon dioxide; leg amputation; wound healing failure; amputation revision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- leg amputation: Patients undergoing below-knee and above ankle amputation for vascular reasons will receive transcutaneous oximetry and transcutaneous carbon dioxide measurement

SUMMARY:
TCOM is a multicentre prospective cohort study in patients undergoing lower limb amputations. Patients will provide oxygen and carbon dioxide measurements in the lower limb for 20 to 30 minutes before their surgery and will be followed up until 6 months after their surgery. The purpose of the TCOM study is to determine the ability of oxygen and carbon dioxide measurements in the legs of patients undergoing lower limb amputation to predict wound healing complications and to determine an optimum cutoff value for both oxygen and carbon dioxide levels beyond which healing complications are likely to occur and a closer amputation level is indicated.

DETAILED DESCRIPTION:
Lower limb amputation is a serious and unfortunate outcome for many patients with vascular disease, especially those with diabetes. It results in significant decreases in all aspects of quality of life. The need for further surgery to revise the amputation to a more proximal level leads to increased potential for serious and life-threatening complications, as well as a decrease in patient morale. From surveys and background literature, it can be estimated that there are approximately 8600 vascular disease-related lower limb amputations in Canada each year. As the epidemic of diabetes continues to unfold and the mean age of the population increases, this number is expected to increase. The results of this study may significantly assist in the surgical and clinical care of this patient population by providing clinicians with a means to assess appropriate lower limb amputation levels.

Further, the modalities of transcutaneous measures may assist in guiding further intervention studies in higher risk patients to improve clinically important outcomes. This study will act in part as a feasibility trial for a randomized controlled trial assessing the efficacy of supplemental oxygen therapy, including hyperbaric oxygen therapy, as a therapeutic tool to increase rates of healing after lower limb amputation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Requires a lower limb amputation between the ankle and knee due to vascular complications
3. Provides written informed consent

Exclusion Criteria:

1. Requires a lower limb amputation for non-vascular reasons, including trauma and cancer
2. Requires primary amputation below the level of the ankle or above the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing below-knee and above-ankle amputations due to vascular complications
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause 30-day mortality and healing failure of the surgical stump | 30 days post-surgery
  Composite of all-cause 30-day mortality and healing failure of the surgical stump at 30 days postoperatively, defined as the need for amputation revision.

SECONDARY OUTCOMES:
6-month all-cause mortality. | 6 months post-surgery
  6-month all-cause mortality
Incidence of re-amputation from 30 days to 6 months post-amputation | 6 months post-surgery
  Incidence of re-amputation from 30 days to 6 months post-amputation
Use of prosthesis for mobilization within 6 months post-amputation | 6 months post-surgery
  Use of prosthesis for mobilization within 6 months post-amputation
Change in health-related quality of life from baseline at 6-months post-amputation | 6 months post-surgery
  Change in health-related quality of life from baseline at 6-months post-amputation, based on the quality of life questionnaire (EuroQoL-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, MD, FRCPC, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada